CLINICAL TRIAL: NCT02172261
Title: Relative Bioavailability of Both BI 10773 and Glimepiride After Co-administration Compared to Multiple Oral Doses of BI 10773 (50 mg q.d.) Alone and a Single Dose of Glimepiride (1 mg) Alone in Healthy Male Volunteers (an Open-label, Randomised, Crossover, Clinical Phase I Study)
Brief Title: Relative Bioavailability of BI 10773 and Glimepiride in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1245.7
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; glimepiride

ARMS (2):
- Sequence ABC (Experimental): 1. Treatment A: BI 10773 once daily from day 1 to 5
  2. Treatment B: BI 10773 and glimepiride once on day 1
  3. Treatment C: Glimepiride once on day 1
  Interventions: Drug: BI 10773; Drug: Glimepiride
- Sequence CAB (Experimental): 1. Treatment C: Glimepiride once on day 1
  2. Treatment A: BI 10773 once daily from day 1 to 5
  3. Treatment B: BI 10773 and glimepiride once on day 1
  Interventions: Drug: BI 10773; Drug: Glimepiride

INTERVENTIONS:
Drug: BI 10773
Drug: Glimepiride

SUMMARY:
The objective was to investigate whether there was a drug-drug interaction between BI 10773 and glimepiride when co-administered. Therefore, the relative bioavailabilities of BI 10773 and glimepiride were determined when both drugs were given in combination compared to multiple oral doses of BI 10773 once daily alone and a single oral dose of glimepiride given alone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
* Age 18 to 50 years (incl.)
* BMI (Body Mass Index) 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP (Blood Pressure, PR (Pulse Rate) and ECG (Electrocardiogram)) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 30 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* Glucose-6-phosphate dehydrogenase deficiency

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) of BI 10773 | up to 5 days
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) of BI 10773 | up to 5 days
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) of glimepiride | up to 4 days
Cmax (maximum measured concentration of the analyte in plasma) of glimepiride | up to 4 days

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) of glimepiride | up to 4 days
tmax (time from dosing to the maximum concentration of the analyte in plasma) of glimepiride | up to 4 days
λz (terminal rate constant in plasma) of glimepiride | up to 4 days
t½ (terminal half-life of the analyte in plasma) of glimepiride | up to 4 days
MRTpo (mean residence time of the analyte in the body after po administration) of glimepiride | up to 4 days
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) of glimepiride | up to 4 days
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) of glimepiride | up to 4 days
tmax,ss (time from last dosing to maximum concentration of the analyte in plasma at steady state over a uniform dosing interval τ) of BI 10773 | up to 5 days
Aet1-t2 (amount of analyte eliminated in urine over the time interval from t1 to t2) of glimepiride | 1 hour pre-dose and 0-2, 2-4, 4-8, 8-12, 12-24 after administration on day 1
fet1-t2 (fraction of analyte excreted unchanged in urine over the time interval from t1 to t2) of glimepiride | 1 hour pre-dose and 0-2, 2-4, 4-8, 8-12, 12-24 after administration on day 1
CLR (renal clearance of the analyte) of glimepiride | 1 hour pre-dose and 0-2, 2-4, 4-8, 8-12, 12-24 after administration on day 1
λz,ss (terminal rate constant of analyte in plasma at steady-state) of BI 10773 | up to 5 days
t½,ss (terminal half-life of analyte in plasma at steady-state) of BI 10773 | up to 5 days
MRTpo,ss (mean residence time of the analyte in the body at steady state after oral administration) of BI 10773 | up to 5 days
CL/F,ss (apparent clearance of the analyte in the plasma after extravascular administration at steady state) of BI 10773 | up to 5 days
Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following extravascular administration) of BI 10773 | up to 5 days
Aet1-t2,ss (amount of analyte eliminated in urine at steady state over a uniform dosing interval τ) of BI 10773 | 1 hour pre-dose and 0-2, 2-4, 4-8, 8-12, 12-24 after administration on day 1 and 5
fet1-t2,ss (fraction of analyte excreted unchanged in urine at steady state over a uniform dosing interval τ) of BI 10773 | 1 hour pre-dose and 0-2, 2-4, 4-8, 8-12, 12-24 after administration on day 1 and 5
CLR,ss (renal clearance of the analyte at steady state) of BI 10773 | 1 hour pre-dose and 0-2, 2-4, 4-8, 8-12, 12-24 after administration on day 1 and 5
UGE0-24 (Urinary glucose excretion of the analyte in urine over the time interval from time zero to 24 h) | 1 hour pre-dose and 0-2, 2-4, 4-8, 8-12, 12-24 after administration on days 1 and 5
Number of patients with abnormal findings in physical examination | Baseline and within 3-14 days after last glimepiride administration
Number of patients with clinically significant changes in vital signs (blood pressure, pulse rate) | Baseline, day 1 and within 3-14 days after last glimepiride administration
Number of patients with abnormal findings in 12-lead ECG (electrocardiogram) | Baseline, day 1 and within 3-14 days after last glimepiride administration
Number of patients with abnormal findings in clinical laboratory tests | Baseline, day 1,4 and within 3-14 days after last glimepiride administration
Number of patients with adverse events | Up to 34 days
Assessment of tolerability by investigator on a 4-point scale | Within 3-14 days after last glimepiride administration
Number of patients with abnormal findings in glucose bedside tests | Pre-dose and 1, 2, 4, 7, 10, 14, 24 hours after glimepiride administration on day 1